CLINICAL TRIAL: NCT01932177
Title: EVESOR: a Phase 1 Trial of Everolimus and Sorafenib to Assess the Impact of Doses and Administration Sequences on Pharmacokinetic and Pharmacodynamic Effects of the Combination
Brief Title: EVESOR: a Phase 1 Trial of Everolimus and Sorafenib
Acronym: EVESOR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-716
Record Dates: First submitted 2013-05-13; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic or Locally Advanced Solid Tumors
Keywords: Everolimus ; Sorafenib ; Phase 1 trial ; Solid tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Schedule A (Active Comparator): Everolimus run-in period followed by continuous administration of everolimus and sorafenib
  Interventions: Drug: Everolimus and sorafenib
- Schedule B (Active Comparator): Sorafenib run-in period followed by continuous administration of everolimus and sorafenib
  Interventions: Drug: Everolimus and sorafenib
- Schedule C (Experimental): Everolimus and sorafenib in alternance
  Interventions: Drug: Everolimus and sorafenib
- Schedule D (Experimental): Continuous administration of everolimus and intermittent administration of sorafenib
  Interventions: Drug: Everolimus and sorafenib

INTERVENTIONS:
Drug: Everolimus and sorafenib — Everolimus will be given alone during a 2 week run-in period before starting sorafenib. Subsequently sorafenib will be administered twice a day while everolimus will be given once a day continuously.
Drug: Everolimus and sorafenib — Sorafenib will be given alone during a 2 week run-in period before starting everolimus. Subsequently sorafenib will be administered twice a day while everolimus will be given once a day continuously.
Drug: Everolimus and sorafenib — Bid sorafenib will be given every other week alternating with 1 week qd everolimus. Doses will be escalated.
Drug: Everolimus and sorafenib — Sorafenib will be given twice a day for 3 days-on 4 days-off while everolimus will be administered continuously on a daily basis. Doses will be escalated.

SUMMARY:
EVESOR multiparameter phase I trial aims at determining the safety of different doses and dosing schedules of everolimus in combination with sorafenib as well as the recommended doses & dosing schedules for phase 2 trials in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
The present phase I trial aims at determining the safety of different doses and dosing schedules of everolimus in combination with sorafenib as well as the recommended doses & dosing schedules for phase 2 trials in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors (breast adenocarcinomas, colorectal adenocarcinomas, renal cell carcinomas, gastric and oesophageal adenocarcinomas, pancreatic cancers, hepatocellular carcinoma, ovarian and Fallopian tube adenocarcinomas, primary peritoneal carcinoma, endometrial and cervix cancers, non-small cell lung carcinoma, melanoma, thyroid carcinomas) resistant or not amenable to standard treatments
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Patients must have assessable primary or metastatic lesion using dynamic contrast enhanced ultrasound
* Patients must be willing to have two tumor biopsies performed (one before study start and one during study treatment), unless medically contraindicated.
* No previous treatment with sorafenib and everolimus. Patients may have been previously treated with one experimental drug: sorafenib or everolimus.
* No other limitation on prior therapy. However, there must be at least a 4 week interval between initiation of study treatment and any prior radiotherapy or systemic therapy, 6 weeks if the last regimen included BCNU or mitomycin C.
* Males and females aged >18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status ≤ 2 (Karnofsky > 70%; see Appendix A).
* Patients must have normal organ and marrow function.
* Patients must be able to swallow medication.
* Pregnancy Testing. Women of childbearing potential are required to have a negative serum pregnancy test within 10-14 days and within 24 hours prior to the first dose of either drug (serum or urine).
* Ability to understand and the willingness to sign a written informed consent document.
* Patient without any legal protection measure and having health coverage.

Exclusion Criteria:

* Previous treatment with sorafenib and everolimus.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus or sorafenib or other agents used in the study.
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible.
* Patients who are taking concurrent medications that are strong inducers/inhibitors of CYP3A4 should be switched to alternative medications to minimize any potential risk. If such patients cannot be switched to alternative medications, they will be ineligible to participate in this study. A list of prohibited CYP3A4 inducers and inhibitors is provided in Appendix D.
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption.
* Patients who are serologically positive for Hepatitis A, B or C, or have other forms of hepatitis or cirrhosis are ineligible, except for patients with hepatocellular carcinoma. Patients with hepatocellular carcinoma with Child Pugh B or C score.
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with everolimus.
* Cardiovascular: Patients with QTc ≥ 470 mSec, as measured by ECG using Bazett's formula for both male and female are ineligible.
* Patients who have not recovered from side effects of previous systemic anticancer therapy to ≤ CTCAE Grade 2 prior to the first dose of combination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Safety (dose limiting toxicities) as well as the recommended doses & dosing schedules for phase 2 trials in adult patients with advanced solid tumors. | Patients will be evaluated for dose limiting toxicities during the first 28-day cycle.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of everolimus in combination with sorafenib | During the first 28-day cycle
  Search for interactions

OTHER OUTCOMES:
Response rate | Every 2 weeks
  Preliminary antitumor activity of everolimus-sorafenib combination
Pharmacodynamic (PD) effects | During the first 28-day cycle
  Pharmacodynamic (PD) effects of everolimus in combination with sorafenib on PI3K-AKT-mTor and RAS-RAF-ERK signaling pathways in tumor and surrogate tissues
PK-PD relationships | During the first 28-day cycle
  Relationships between PK and PD effects measured in tumor and surrogate tissues

CONTACTS AND LOCATIONS:
Overall Officials: BENOIT YOU, MD PhD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Puszkiel A, You B, Payen L, Lopez J, Guitton J, Rousset P, Fontaine J, Peron J, Maillet D, Tartas S, Bonnin N, Trillet-Lenoir V, Colomban O, Augu-Denechere D, Freyer G, Tod M. A PK-PD model linking biomarker dynamics to progression-free survival in patients treated with everolimus and sorafenib combination therapy, EVESOR phase I trial. Cancer Chemother Pharmacol. 2023 May;91(5):413-425. doi: 10.1007/s00280-023-04520-z. Epub 2023 Apr 3. PMID 37010549
- [Derived] Varnier R, Puszkiel A, Tod M, Calattini S, Payen L, Lopez J, Guitton J, Schwiertz V, Fontaine J, Peron J, Maillet D, Tartas S, Bonnin N, Colomban O, Augu-Denechere D, Freyer G, You B. Clinical results of the EVESOR trial, a multiparameter phase I trial of everolimus and sorafenib combination in solid tumors. Cancer Chemother Pharmacol. 2023 May;91(5):361-373. doi: 10.1007/s00280-023-04508-9. Epub 2023 Feb 25. PMID 36840749
- [Derived] El-Madani M, Colomban O, Tod M, Maillet D, Peron J, Rodriguez-Lafrasse C, Badary OA, Valette PJ, Lefort T, Cassier P, El-Shenawy SM, El-Demerdash E, Hommel-Fontaine J, Guitton J, Gagnieu MC, Ibrahim BM, Barrois C, Freyer G, You B. EVESOR, a model-based, multiparameter, Phase I trial to optimize the benefit/toxicity ratio of everolimus and sorafenib. Future Oncol. 2017 Apr;13(8):679-693. doi: 10.2217/fon-2016-0357. Epub 2017 Jan 12. PMID 28076966